CLINICAL TRIAL: NCT06078098
Title: Multicenter, Nationwide, Observational, Retrospective and Prospective Study Based on the Development of a Autoimmune Hepatitis Patient's Database Linked to a Biological Sample Storage
Brief Title: Development of a Autoimmune Hepatitis Patient's Database Linked to a Biological Sample Storage
Acronym: AIH Database
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: AIH Database
Record Dates: First submitted 2023-03-31; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Autoimmune Hepatitis; Liver Disorder
Keywords: Autoimmune Hepatitis; National Database; Liver; Epidemiology
MeSH Terms: conditions — Hepatitis, Autoimmune; Digestive System Diseases | interventions — Clinical Laboratory Information Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 11 Years
Biospecimen Retention: Samples With DNA — The collection of biological samples is facultative. Biological samples are collected at time of recruitment and on a yearly basis (for blood, urine and stools). The collection of liver tissue depends on the specific procedures (liver biopsy) which are performed based on clinical needs.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AIH patients: AIH population in Italy aged at least 1 year
  Interventions: Other: Clinical Information

INTERVENTIONS:
Other: Clinical Information — We will recruit AIH patients and collect important clinical information and laboratory investigation, together with biological samples.
  Other Names: Laboratory information; Biological samples

SUMMARY:
Autoimmune Hepatitis (AIH) is chronic fibroinflammatory disease of the liver characterized by chronic, relapsing liver inflammation, and a risk for progression to liver failure and need for liver transplantation. No AIH-specific registry does exist in Italy, so that the actual epidemiology of the disease in the country is unknown.

This is an observational, retrospective and prospective, multicenter study evaluating incidence, prevalence and disease course of AIH in subjects > 1 years old in Italy.

DETAILED DESCRIPTION:
Autoimmune Hepatitis (AIH) is a chronic fibroinflammatory disease of the liver characterized by chronic, relapsing inflammation, and a risk for progression to liver failure and development of hepatocellular cancer. Both children and adults are affected. A significant fraction of patients with AIH has a diminished life expectancy, despite treatment. Around 80% of patients respond to current therapies, but their quality of life and health is hugely impaired by side effects. The remaining proportion of patients (the difficult-to-treat category) do not respond to treatment and progress to liver cirrhosis and its complications; thus, timely identification of these individuals is a key aspect of epidemiological research in AIH.Taken together and combined with patients' debilitating quality of life issues, these data highlight the considerable disease burden and clinical impact of AIH on patients' outcomes.

Most epidemiological studies on AIH are retrospective case series based on tertiary referral series with relevant selection biases. Population-based studies, that include all cases in a defined geographical area, provide more accurate estimates of incidence, survival and mortality rate for the individual with AIH. Typically, multiple case-finding approaches have been used, including surveys, laboratory reports, liver histology databases, transplant registries, and death certificates. Only few population-based studies have been performed and limit the research population to a few dozen patients, reporting incidence rates ranging from 1.07 to 1.9 per 100,000 inhabitants. Reported point prevalence is 16.9 per 100,000.

To the investigators knowledge, there have been no epidemiologic studies in AIH carried out in Italy.

The investigators aim to develop a national registry on this rare disease to describe incidence and prevalence of AIH in Italy; identify and define distinct phenotypes and sub-phenotypes of AIH patients; identify factors influencing the progression of AIH and affecting mortality; assess safety and long-term efficacy of novel therapies.

This is a multicentre, nationwide, observational and prospective study based on the development of a patient's database linked to a biological sample storage. The enrollment period will cover 120 months to include the required number of patients. Based on litteraure, the estimated prevalence of AIH in Italy ranges from 6,000 to 15,000. Based on this, the investigators estimate to enroll approximately 10,000 patients. The minimum follow-up time will be 1 year.

ELIGIBILITY:
Inclusion Criteria:

* All AIH patients living in Italy and aged at least 1 year can be included in the database.
* Willing and able to give informed consent prior to any study specific procedure being
* Diagnosis of AIH according to the most recent published guidelines (EASL)

Exclusion Criteria:

* Subject unwilling to participate at the study

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Italian AIH patients (diagnosis of AIH according to the most recent published guidelines EASL) aged at least 1 year
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2034-03-29 (Estimated); Study Completion 2034-03-29 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Normalization of AST and ALT <1 x upper limit of normal (ULN)) and normal IgG levels within 6 months | Overall duration of the study (11 years)
  Number of participants with Normalization of AST and ALT <1 x upper limit of normal (ULN)) and normal IgG levels within 6 monthswithin 6 months
Number of participants with lack of biochemical response | Overall duration of the study (11 years)
  Number of participants with lack of biochemical response
Number of participants with <50% decrease of AST and ALT within 4 weeks after initiation of treatment | Overall duration of the study (11 years)
  Number of participants with <50% decrease of AST and ALT within 4 weeks after initiation of treatment
Number of participants with Hepatitis Activity Index <4/18 | Overall duration of the study (11 years)
  Number of participants with Hepatitis Activity Index <4/18
Intolerance to treatment | Overall duration of the study (11 years)
  Any adverse event possibly related to treatment as assessed by the treating physician leading to potential discontinuation of the drug
Deep biochemical remissionof disease progression | Overall duration of the study (11 years)
  ALT less than 50% ULN and IgG<12g/l
Relapse | Overall duration of the study (11 years)
  An increase in serum ALT levels above three times the ULN and/or an increase in serum IgG levels to more than 20 g/l
Number of participants with An increase in serum ALT levels above ULN on at least two occasions with an interval of 4 weeks | Overall duration of the study (11 years)
  Number of participants with An increase in serum ALT levels above ULN on at least two occasions with an interval of 4 weeks, with or without concomitant clinical symptoms and reinstitution of drug therapy after exclusion of other plausible causes for the elevated serum ALT
Number of participants with variceal bleeding requiring hospital admission | Overall duration of the study (11 years)
  Number of participants with variceal bleeding requiring hospital admission
Number of participants with first evidence of ascites requiring hospital admission | Overall duration of the study (11 years)
  Number of participants with first evidence of ascites requiring hospital admission
Number of participants with hepatic encephalopathy requiring hospital admission | Overall duration of the study (11 years)
  Number of participants with hepatic encephalopathy requiring hospital admission
Number of participants with serum bilirubin levels > 1.0 mg/dl on more than one consecutive sample | Overall duration of the study (11 years)
  Number of participants with serum bilirubin levels > 1.0 mg/dl on more than one consecutive sample
Number of participants with platelet count < 150.000/mm3 on more than one consecutive sample | Overall duration of the study (11 years)
  Number of participants with platelet count < 150.000/mm3 on more than one consecutive sample
Number of participants with albumin levels < 3.5 mg/dL on more than one consecutive sample | Overall duration of the study (11 years)
  Number of participants with albumin levels < 3.5 mg/dL on more than one consecutive sample

SECONDARY OUTCOMES:
Liver stiffness | Overall duration of the study (11 years)
  Liver stiffness by fibroscan
Number of participants achieving HAI score < 4 at follow-up biopsies | Overall duration of the study (11 years)
  Number of participants achieving HAI score < 4 at follow-up biopsies
The time from the diagnosis of AIH to an event | Overall duration of the study (11 years)
  Date of diagnosis of AIH: Defined as the date of the diagnostic liver biopsy, or the date of the first abnormal AST or ALT, or the date of starting therapy in those cases that did not perform a liver biopsy at baseline but fulfilled diagnostic criteria for the disease. Events: Defined as follows: (1) death from a liver-related cause, meaning liver failure, variceal hemorrhage, or HCC; (2) Liver Transplantation for AIH

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS San Gerardo dei Tintori, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heneghan MA, Yeoman AD, Verma S, Smith AD, Longhi MS. Autoimmune hepatitis. Lancet. 2013 Oct 26;382(9902):1433-44. doi: 10.1016/S0140-6736(12)62163-1. Epub 2013 Jun 14. PMID 23768844
- [Background] Sharma R, Verna EC, Soderling J, Roelstraete B, Hagstrom H, Ludvigsson JF. Increased Mortality Risk in Autoimmune Hepatitis: A Nationwide Population-Based Cohort Study With Histopathology. Clin Gastroenterol Hepatol. 2021 Dec;19(12):2636-2647.e13. doi: 10.1016/j.cgh.2020.10.006. Epub 2020 Oct 14. PMID 33065308
- [Background] Mack CL, Adams D, Assis DN, Kerkar N, Manns MP, Mayo MJ, Vierling JM, Alsawas M, Murad MH, Czaja AJ. Diagnosis and Management of Autoimmune Hepatitis in Adults and Children: 2019 Practice Guidance and Guidelines From the American Association for the Study of Liver Diseases. Hepatology. 2020 Aug;72(2):671-722. doi: 10.1002/hep.31065. Epub 2020 May 12. No abstract available. PMID 31863477
- [Background] Wong LL, Fisher HF, Stocken DD, Rice S, Khanna A, Heneghan MA, Oo YH, Mells G, Kendrick S, Dyson JK, Jones DEJ; UK-AIH Consortium. The Impact of Autoimmune Hepatitis and Its Treatment on Health Utility. Hepatology. 2018 Oct;68(4):1487-1497. doi: 10.1002/hep.30031. PMID 29663477
- [Background] Pape S, Snijders RJALM, Gevers TJG, Chazouilleres O, Dalekos GN, Hirschfield GM, Lenzi M, Trauner M, Manns MP, Vierling JM, Montano-Loza AJ, Lohse AW, Schramm C, Drenth JPH, Heneghan MA; International Autoimmune Hepatitis Group (IAIHG) collaborators(double dagger). Systematic review of response criteria and endpoints in autoimmune hepatitis by the International Autoimmune Hepatitis Group. J Hepatol. 2022 Apr;76(4):841-849. doi: 10.1016/j.jhep.2021.12.041. Epub 2022 Jan 20. PMID 35066089
- [Background] Heneghan MA, Shumbayawonda E, Dennis A, Ahmed RZ, Rahim MN, Ney M, Smith L, Kelly M, Banerjee R, Culver EL. Quantitative magnetic resonance imaging to aid clinical decision making in autoimmune hepatitis. EClinicalMedicine. 2022 Mar 21;46:101325. doi: 10.1016/j.eclinm.2022.101325. eCollection 2022 Apr. PMID 35340625
- [Background] van Gerven NM, Verwer BJ, Witte BI, van Hoek B, Coenraad MJ, van Erpecum KJ, Beuers U, van Buuren HR, de Man RA, Drenth JP, den Ouden JW, Verdonk RC, Koek GH, Brouwer JT, Guichelaar MM, Mulder CJ, van Nieuwkerk KM, Bouma G; Dutch Autoimmune Hepatitis Working Group. Relapse is almost universal after withdrawal of immunosuppressive medication in patients with autoimmune hepatitis in remission. J Hepatol. 2013 Jan;58(1):141-7. doi: 10.1016/j.jhep.2012.09.009. Epub 2012 Sep 16. PMID 22989569